CLINICAL TRIAL: NCT02852447
Title: The Effect of Surgery for Non Endometriosic Ovarian Cysts on Ovarian Reserve : A Prospective Study
Brief Title: The Effect of Surgery for Non Endometriosic Ovarian Cysts on Ovarian Reserve
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Laura Costa-Canals, MD, Corporacion Parc Tauli
Other Study IDs: CPT-GINE-2016
Record Dates: First submitted 2016-07-01; First posted 2016-08-02 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Antimullerian Hormone; Ovarian Cysts; Antral Follicle Count
MeSH Terms: conditions — Ovarian Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood

SUMMARY:
The main objective is to evaluate the ovarian reserve after laparoscopic cystectomy.

The secondary objective is the analysis of predictors of change in the ovarian reserve after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients with non endometriosis ovarian cysts
* Age between 15-40 years
* Regulars menses
* Signed informed consent

Exclusion Criteria:

* Patients with Previous surgery,
* Patients with infertility,
* Patients with endometriosis or
* Patients with suspicious of malignance

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with bening ovarian cyst and requiring surgical removal
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
differences in the ovarian reserve before and after surgery by Antimullerian Hormone | 3 months
differences in the ovarian reserve before and after surgery by Antral Follicle Count | 3 months

SECONDARY OUTCOMES:
Ovarian Size (mm) | 3 months
Time of surgery (minutes) | 3 months
Age (years) | 3 months
BMI in kg/m2 | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Corporació Sanitària Parc Tauli, Sabadell, Barcelona, Spain